CLINICAL TRIAL: NCT04386928
Title: Allogeneic Stem Cell Transplantation (ALLO-SCT) in Elderly: 17-years Retrospective GITMO Survey
Brief Title: ALLO-SCT in Elderly Patients With Hematological Disease
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Trapianto di Midollo Osseo (Other)
Collaborators: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Sponsor
Other Study IDs: GITMO-AlloElderly
Record Dates: First submitted 2020-05-05; First posted 2020-05-13 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Hematologic Diseases; Stem Cell Transplant Complications
Keywords: Allogeneic stem cell transplantation; Elderly; Retrospective survey; GITMO; Hematological disease
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly patients with hematological disease: older than 60 years who received hematopoietic stem cell transplantation (HSCT)

SUMMARY:
Retrospective, observational, multicentre, spontaneous, non-interventional study This study will evaluate all consecutive patients older than 60 years who received hematopoietic stem cell transplantation (HSCT) between 1st January 2000 and 31st December 2017.

DETAILED DESCRIPTION:
The age of patients' population is increasing every year, as the life expectancy. Thus, the incidence and prevalence of hematological cancers is increasing. In particular, acute leukemias and myelodysplastic syndromes are the most frequent diseases of the hematopoietic system. Allogeneic stem cell transplantation (allo-SCT) is the main therapeutic options for these diseases, and the number of allo-SCTs in the elderly is currently in progressive growth. This is partially due to the improvement of the allo-SCT procedure over the years, with the amelioration of donor selection, Human Leukocyte Antigen typing, graft versus host disease (GVHD) and infections prophylaxis and treatment.

Nevertheless, there is still an unmet clinical need, represented by the lack of extensively and detailed outcome analysis of elderly patients addressed to allo-SCT. With this aim, the investigators planned this retrospective analysis of allo-SCTs in patients older than 60 years, within the Gruppo Italiano Trapianti di Midollo Osseo transplant activity of the last 17 years. This study will help us in designing future prospective trials, including a comprehensive geriatric assessment of frailty, in order to address to allo-SCT those elderly who have the highest probability to achieve the best long term outcome with the lowest transplant-related mortality and morbidity.

For patients submitted to more than one transplant, the first transplant will be considered only and the record of these patients will be derived from the Gruppo Italiano Trapianti di Midollo Osseo database and the European group for Blood and Marrow Transplantation database (Promise), where all the transplant activity is regularly recorded.

Primary objective is description of the patients' population. This endpoint will particularly focus on the changing, over the years, of the clinical and hematological characteristics of elderly patients submitted to allo-SCT.

Secondary objectives are: description of the transplants' characteristics, such as the conditioning regimens and the GVHD prophylaxis, description of acute and chronic graft versus host disease (GVHD) incidence and treatment, description of overall survival (OS), disease-free survival (DFS), transplant related mortality (TRM) and relapse risk (RR).

The sample size includes all the transplants recorded in the Gruppo Italiano Trapianti di Midollo Osseo and European group for Blood and Marrow Transplantation database. The statistical analysis will be descriptive, so the investigators don't need to calculate a sample size for the study. This analysis will include:

* full description of patients and transplant characteristics. In this area, a specific focus will be done on the pre-transplant comorbidity index, according to the most commonly published risk-scores.
* focus on acute and chronic GVHD incidence and treatment.
* outcome description, with a focus on: Overall Survival, Disease Free Survival), Transplant Related Mortality, relapse risk.

These outcome measures will be assessed at 1, 2 and 5 years from allo-SCT. The analysis of the continuous and categorical variables will take place according to the criteria of the descriptive statistics, including mean, median, standard deviation, range, minimum values and maximum values for the continuous variables, absolute and relative values for the categorical variables. For the comparison of continuous and categorical variables, parametric and non-parametric statistical tests will be applied (Chi-square test, Fisher exact test and rank correlation coefficient of Spearman).

This trial is being organized under the auspices of the Gruppo Italiano Trapianti di Midollo Osseo that involves the principal Centres active in transplantation of any kind of hematopoietic stem cells (HSCT) in Italy.

The study will be conducted according to the principles of Good Clinical Practice, the current Italian and European laws and regulations, in agreement with the declaration of Helsinki. The protocol has been written and the study will be conducted according to the The International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) Harmonized Tripartite Guideline for Good Clinical Practice, issued by the European Union. The responsible Local Ethical Committee approval must be obtained before starting the trial. A copy of the patient informed consent form must be submitted to the appropriate authority or committee, together with the protocol for written approval. Written approval of the protocol and informed consent by the responsible and appropriate authority or committee must be obtained prior to recruitment of patients to the study.

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic transplantation from 2000 to 2017 (for patients submitted to more than one transplant, only the first transplant will be considered)
* Informed consent

Exclusion Criteria:

* Absence of informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enrol patients older than 60 years who received hematopoietic stem cell transplantation (HSCT) between 1st January 2000 and 31st December 2017.
Sampling Method: Probability Sample
Enrollment: 1996 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | These outcome measures will be assessed at 5 years from allo-SCT.
  is defined as the time from transplant to the date of death due to any cause or to the last date the patient was known to be alive (censored observation) or to the date of the data cut-off for final analysis
Disease Free Survival (DFS) | These outcome measures will be assessed at 5 years from transplant
  DFS is defined as the probability of being alive free of disease at any point in time.
Transplant Related Mortality (TRM) | These outcome measures will be assessed at 5 years from transplant
  TRM was defined as death due to any transplantation-related cause other than disease relapse
Relapse risk (RR) | These outcome measures will be assessed at 5 years from transplant.
  The relative risk (RR) or risk ratio is the ratio of the probability of an outcome in an exposed group to the probability of an outcome in an unexposed group.

SECONDARY OUTCOMES:
Acute Graft-versus-Host Disease | These outcome measures will be assessed at 100 days from transplant
  cumulative incidence of acute GvHD (grade II-IV)
Chronic Graft-versus-Host Disease | These outcome measures will be assessed at 5 years from transplant
  cumulative incidence and severity of chronic graft-versus-host disease

CONTACTS AND LOCATIONS:
Overall Officials: Michele Malagola, MD, Principal Investigator — ASST Spedali Civili di Brescia
Locations (29):
- Italy (29):
  - Azienda Ospedaliero-Universitaria Ospedali Riuniti, Ancona
  - Ospedale Mazzoni, Ascoli Piceno
  - Policlinico di Bari-Ematologia con trapianti, Bari
  - Ospedale San Orsola, Bologna
  - Ospedale Regionale Generale- Divisione Ematologia, Bolzano
  - ASST Spedali Civili, Brescia
  - CTMO PO "Businco" A.O. "G. Brotzu", Cagliari
  - Azienda Ospedaliera di Careggi, Florence
  - Osp. Card. Panico, Lecce
  - Ospedale dell'Angelo, Mestre
  - Ospedale Maggiore - Policlinico, Milan
  - Ospedale Niguarda Ca' Grande, Milan
  - Ospedale San Raffaele, Milan
  - Divisione Ematologia - Azienda Ospedaliera Universitaria - Policlinico -, Modena
  - ASST Ospedale S. Gerardo de' i Tintori - Università degli Studi di Milano, Monza
  - A.O.U. San Luigi Gonzaga, Orbassano
  - IRCCS Policlinico S. Matteo, Pavia
  - Ospedale Civile, Pescara
  - Ospedale G. Da Saliceto di Piacenza, Piacenza
  - Centro Unico Regionale Trapianti di Midollo Osseo - Ospedale Bianchi-Melacino-Morelli, Reggio Calabria
  - Divisione di Ematologia - Istituto di Semeiotica Medica - Policlinico A. Gemelli, Roma
  - Policlinico Umberto I, Roma
  - U.O. di Ematologia e Trapianti di Midollo Osseo - Azienda Osp. S. Camillo-Forlanini / Padiglione Morgagni, Roma
  - AOU S. Giovanni di Dio e Ruggi d'Aragona, Salerno
  - Ematologia e Centro Trapianti Midollo Osseo - Ospedale IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Ospedale Moscati, Taranto
  - A.O.U. Citta della Salute e della Scienza, Torino
  - Clinica Ematologica - Policlinico Universitario, Udine
  - Ospedale S. Bortolo-Divisione Ematologia, Vicenza